CLINICAL TRIAL: NCT02589288
Title: Adductor Canal Block: Continuous Infusion Versus Automatic Intermittent Bolus For Postoperative Analgesia After Day-Case Anterior Cruciate Ligament Reconstruction
Brief Title: Adductor Canal Block: Continuous Infusion Versus Automatic Intermittent Bolus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, MD, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOGPGC09
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Injury of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Infusion (Active Comparator): Patients receive a postoperative continuous infusion of Ropivacaine 0,2% at 6 ml/h and 4 ml PCA bolus, lockout 20 minutes via electronic infusion pump (Micrel device, Greece).
  Interventions: Procedure: Continuous Infusion of ropivacaine 0.2%
- Automatic Intermittent Bolus (Experimental): Patients receive a postoperative Automatic Intermittent Bolus of 6 ml Ropivacaine 0,2% and 4 ml PCA bolus, lockout 20 minutes every hour via electronic infusion pump (Micrel device, Greece).
  Interventions: Procedure: Automatic Intermittent Bolus of ropivacaine 0.2%

INTERVENTIONS:
Procedure: Continuous Infusion of ropivacaine 0.2% — Postoperative continuous infusion of Ropivacaine 0,2% at 6 ml/h and 4 ml PCA bolus, lockout 20 minutes via electronic infusion pump (Micrel device, Greece).
  Other Names: naropine 0.2%
  Arms: Continuous Infusion
Procedure: Automatic Intermittent Bolus of ropivacaine 0.2% — Postoperative Automatic Intermittent Bolus of 6 ml Ropivacaine 0,2% every hour and 4 ml PCA bolus, lockout 20 minutes via electronic infusion pump (Micrel device, Greece).
  Arms: Automatic Intermittent Bolus

SUMMARY:
The aim of this prospective, randomized , blinded study is to compare two different infusion techniques (continuous VS intermittent automatic bolus) to assess the effects of postoperative analgesia after Day-Case anterior cruciate ligament (ACL) reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old
* American society of anesthesiology (ASA) physical status I-II
* Signed informed consensus

Exclusion Criteria:

* ASA >II
* Unstable neurological disease
* Diabetic mellitus (DM) type I-II
* Allergy to used drugs
* Opioid chronic treatment
* Consensus refusal or not valid
* Anticoagulant therapy
* Postoperative intensive care required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
NRS Score | 72h postoperative
  Evaluation of numeric rating score (NRS) in patient with automatic intermittent bolus of Ropivacaine 0,2% instead of classic continuous perfusion

SECONDARY OUTCOMES:
Up and Go test | 72h postoperative
  "up and go" test: time need to get up from a chair, walk for 3 meters, and come back to seat down on the chair
Opioids request | 72h postoperative
  Opioids consumption will be recorded throughout 72 postoperative hours
Local anesthetic consumption | 72h postoperative
  Evaluation of local anesthesia consumption every 6h in first 72 postoperative hours.
10mt walk test | 72h postoperative
  time need to walk 10 meters

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Cappelleri, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Istituto ortopedico Gaetano Pini, Milan, Italy